CLINICAL TRIAL: NCT01533818
Title: Community Based Management of Fast Breathing in Infants Aged < 60 Days: A Double-Blind, Randomized Placebo-Controlled Trial in Low-income Settlements of Karachi
Brief Title: Community Based Management of Fast Breathing in Infants Aged < 60 Days in Low-income Settlements of Karachi
Acronym: MAT-YI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped by DSMB based on high treatment failure rate in placebo compared to active drug.
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Shiyam Sunder Tikmani, Research Supervisor, Aga Khan University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1979-CHS-ERC-11
Record Dates: First submitted 2012-02-13; First posted 2012-02-15 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Fast Breathing in Young Infants
Keywords: Fast breathing; Young infants; Management; Amoxicillin; Placebo
MeSH Terms: conditions — Hyperventilation | interventions — Amoxicillin; High Fructose Corn Syrup

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin (Active Comparator): This is an active intervention
  Interventions: Drug: Amoxicillin
- Sugar Syrup (Placebo Comparator)
  Interventions: Drug: Sugar Syrup

INTERVENTIONS:
Drug: Amoxicillin — 80-100 mg/kg/day in 2 divided doses for 7 days
  For convenience dose divided into six weight bands Table 2: Dose of amoxicillin Weight band Amount per dose Daily dose Lower Limit (mg or units /kg/d) Upper Limit (mg or units /kg/d) Amoxicillin - desired range 75-100 mg/kg/day (25mg/ml (125mg/5ml); twice daily orally)* 1.8-1.9 kg 3.0 ml 150 mg 75.4 100.0 2.0-2.4 kg 4.0 ml 200 mg 80.3 100.0 2.5-2.9 kg 5.0 ml 250 mg 83.6 100.0 3.0-3.9 kg 6.0 ml 300 mg 75.2 100.0 4.0-4.9 kg 8.0 ml 400 mg 80.2 100.0 5.0-5.9 kg 10.0 ml 500 mg 83.5 100.0
  Arms: Amoxicillin
Drug: Sugar Syrup — It will be given 2 times/day for 7 days
  Arms: Sugar Syrup

SUMMARY:
The aim of the study is to determine optimal management of isolated fast breathing in young infants in a trial design conducted in primary care settings.

The investigators hypothesized that proportion of infants who fail therapy will be 4% in each group. A 6% or less difference in failure rate will be considered equivalent.

DETAILED DESCRIPTION:
The management of isolated fast breathing is therefore unknown and our experience suggests that these infants could perhaps be managed without antibiotics. Widespread application of the WHO clinical algorithm could therefore result in the referral of as many as 13.7% (135.7 per 1000 live births) of all infants for isolated fast breathing, the vast majority of these unnecessarily, and exposing infants to a high risk of nosocomial sepsis and hospital mortality in addition to over-burdening health resources.

ELIGIBILITY:
Inclusion Criteria

* Young infant (0-59 days of age)
* Fast breathing i.e., respiratory rate ≥60 breaths/min
* O2 Saturation ≥90%
* Resident of catchment area (to ensure complaint and follow up)
* Refused hospitalization and investigations
* Informed consent is provided by a parent (or legal guardian).

Exclusion Criteria:

* Preterm infants (born <37 weeks)
* Presence of audible murmur
* Any concurrent signs of severe infection:
* not feeding well
* movement only when stimulated
* severe chest in-drawing
* axillary temperature ≥38.0oC or ≤35.5oC
* Any sign of being critically ill (Cyanosis, bulging fontanel, unable to feed, unable to cry, apnoea, convulsions, unconscious, persistent vomiting)
* Weight <1800gm at the time of presentation
* Major congenital malformations or suspected chromosomal abnormalities
* Hospitalization for illness in the last two weeks
* Previous inclusion in the study

Max Age: 59 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 963 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Treatment failure | Day 8 of enrollemnt
  1. O2 sat <90% on Day 2 or any time until Day 7.
  2. Clinical deterioration: emergence of any sign of being critically ill or severe infection at any time after randomization (as defined in exclusion criteria)
  3. Development of serious adverse effect of the study antibiotics (death, organ failure, anaphylactic reaction, severe diarrhoea, disseminated and severe rash).
  4. Hospitalization any time after admission in the study.
  5. Death anytime within day 1-7 of enrolment

SECONDARY OUTCOMES:
Compliance to treatment | 80% of total dosage
  To label as per protocol infant should receive 100% (4 doses) of doses in first 2 days followed by 70% (7 doses) of doses from day 3 to day 8.
Proportion of infants relapse | No treatment failure by day 8 and signs of sepsis or fast breathing between day 8-14

CONTACTS AND LOCATIONS:
Overall Officials: Shiyam Sunder P Tikmani, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Primary Health Centers, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Tikmani SS, Muhammad AA, Shafiq Y, Shah S, Kumar N, Ahmed I, Azam I, Pasha O, Zaidi AK. Ambulatory Treatment of Fast Breathing in Young Infants Aged <60 Days: A Double-Blind, Randomized, Placebo-Controlled Equivalence Trial in Low-Income Settlements of Karachi. Clin Infect Dis. 2017 Jan 15;64(2):184-189. doi: 10.1093/cid/ciw690. Epub 2016 Oct 19. PMID 27941119
- See also: Related Info — http://www.aku.edu